CLINICAL TRIAL: NCT06565091
Title: Development Clinical Investigation for a Multifunction Ophthalmic Measurement Device
Brief Title: Clinical Investigation for a Multifunction Ophthalmic Measurement Device
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Essilor International (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: WS10339; 2023-A01481-44 (Other: Agence Nationale de Sécurité du Médicament et des produits de santé (ANSM) - France)
Record Dates: First submitted 2024-08-19; First posted 2024-08-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Accommodation Disorder; Keratoconus; Dry Eye; Refractive Errors; Accommodative Fatigue; Accommodative Inertia; Aberration, Corneal Wavefront
MeSH Terms: conditions — Keratoconus; Dry Eye Syndromes; Refractive Errors; Corneal Wavefront Aberration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multifonction Ophtalmic Measuring Device (Experimental): Parameters and images of the anterior and posterior chambers of the human eye
  Interventions: Device: Measurements of physiological parameters of the anterior chamber; Device: Measurements of the Axial biometry

INTERVENTIONS:
Device: Measurements of physiological parameters of the anterior chamber — Acquisition by the investigational device
Device: Measurements of the Axial biometry — Acquisition by the investigational device

SUMMARY:
The purpose of this clinical investigation is to evaluate the clinical utility of a multifunctional measuring device for Ophtalmology.

The results of this clinical investigation will be used to refine and validate the device design.

378 participants total will be included in the trial, each having only one visit at the investigation center.

DETAILED DESCRIPTION:
The objectives of this clinical investigation are:

* Develop the device in clinical conditions (refine the intensity and gain of the light sources and the acquisition time of the cameras and photodiodes, in order to cover the targeted population).
* Evaluate the safety and clinical performance and/or effectiveness of the medical device and determine whether the system is suitable for the purposes and populations for which it is intended.

ELIGIBILITY:
Inclusion Criteria:

Adults ≥ 18 years old and Healthy children* ≥ 4 years and <18 of age.

Participants initially coming to the center for a routine consultation

Participants who are affiliated to a social security scheme or beneficiaries of such a scheme (L. 1121-8-1 of the Public Health Code of "Code de Santé Publique"),

Participants able to sit upright in front of the investigational device.

Inclusion Criteria* (for Healthy children):

Healthy children ≥ 4 years and <18 of age. The parents must have consented to their child's participation.

Children who are affiliated to parent's social security scheme or beneficiaries of such a scheme (L. 1121-8-1 of the Public Health Code of "Code de Santé Publique")

Children initially coming to the center for a routine consultation

Children able to sit upright in front of the instrument.

Exclusion Criteria:

Participants with implanted electronic medical device such as pacemaker, insulin pump, cochlear implant, electrostimulator or hearing aid,

Participants not able to sit upright in front of the instrument or subjects with forehead or chin injuries which prevent the head from being supported on the forehead / chin rest.

Participants who are deprived of their liberty by judicial or administrative decision and persons hospitalized without their consent (Article L. 1121-6 of "Code de Santé Publique"),

Participants who are subject to a legal protection measure (curatorship, guardianship, safeguard of justice ...) or unable to express their consent (Article L1121-8 of "Code de Santé Publique"),

Participants who are not affiliated to a social security scheme or beneficiaries of such a scheme (L. 1121-8-1 of the Public Health Code of "Code de Santé Publique"),

Participants under exclusion period from another investigation,

Women who are pregnant or breastfeeding women; (Article L1121-5 of "Code de Santé Publique"). No additional risk had been identified for pregnant woman in participating in the investigation. Nevertheless, pregnancy induces ocular changes: in case of AE, the causality with the device or with pregnancy may be difficult to establish, justifying the non-inclusion of this population.

Participants with neurologic disorder, particularly epileptic or sensory motor troubles,

Participants with history of recent ocular surgeries (including refractive surgery less than 2 weeks),

Participants who are ESSILOR International/ESSILOR Luxottica employees,

Participants with monophthalmia,

Participants with obvious fixation disorder, strabismus, or nystagmus,

For tonometry measurements: subjects who have: Edematous/ulcerated cornea, following keratoplasty or ocular surgery, following penetrating trauma, severe Keratoconus with risk of hydrops and in case of retinal detachment. Anterior and posterior chamber sulcus IOL, intrastromal rings or lens (type Kamra).

Participants with pupil < 2 mm,

Participants who are with spherical equivalent refraction out of the range -20.00 to + 20.00 D (frontofocometer measurement),

Participants with an astigmatism greater than 8.00 D (<8.00 D) (frontofocometer measurement),

Participants with corneal power out of the range [35-55D],

Participants with axial length out of the range [18-34 mm],

Participants with Intraocular pressure out of [7-50 mm Hg] range,

Participants to a previous phase of this clinical investigation.

Exclusion Criteria (for Healthy children):

Children with neurologic disorders, particularly epileptic or sensory motor troubles,

Children with history of recent ocular surgeries (including refractive surgery less than two weeks)

Children with monophthalmia,

Children with obvious fixation disorder, strabismus, or nystagmus,

Children with pupil < 2 mm

Children with a spherical equivalent refraction out of the range [-20.00 to + 20.00 D] (frontofocometer measurement),

Children with an astigmatism higher than 8.00 D (>8.00 D)

Children with axial length out of the range [18-34 mm]

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 378 (Estimated)
Dates: Start 2024-06-10 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Relative frequency of successful acquisition for each measurement of the investigational device | One day (measurements are taken during the single visit)

CONTACTS AND LOCATIONS:
Overall Officials: François LE GUYADER, Dr, Principal Investigator — WEST OPHTA
Locations (1):
- West Ophta, Rennes, France